CLINICAL TRIAL: NCT02573701
Title: Comparative Study of Recommended Treatment for Schizophrenia Guideline Treatment vs Treatment as Usual in Child Psychiatric Hospital: Effect on Adherence, Efficacy on Symptoms, and Global Function
Brief Title: Guideline vs Usual Treatment in Schizophrenic Adolescents
Acronym: ACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Psiquiatrico Infantil Dr. Juan N. Navarro, Mexico (Other Government)
Responsible Party: Principal Investigator, Rosa E. Ulloa, Investigator in Medical Sciences, Hospital Psiquiatrico Infantil Dr. Juan N. Navarro, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: II3/02/0811
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Adolescents; Treatment; Guidelines
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Exercise; Population Groups; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Guideline treatment (Experimental): Participants will receive the Guideline Treatment (risperidone, administered orally) plus Behavioral Intervention: "psychosocial treatment" included "psychoeducation" "social skills" "healthy life style habits" "exercise in group"
  Interventions: Drug: Guideline treatment (Risperidone, administered orally); Behavioral: "Psychosocial treatment"
- 2 Treatment as Usual (Active Comparator): Participants will receive the Treatment as Usual (atypical antipsychotic) plus psychosocial treatment decided by clinician
  Interventions: Drug: Treatment as Usual (any other antipsychotic)

INTERVENTIONS:
Drug: Guideline treatment (Risperidone, administered orally) — Participants will receive the Guideline Treatment (risperidone, administered orally) plus Behavioral Intervention: "psychosocial treatment" included "psychoeducation" "social skills" "healthy life style habits" "exercise in group"
  Other Names: Atypical antipsychotic
  Arms: 1 Guideline treatment
Behavioral: "Psychosocial treatment" — Participants will receive the Guideline Treatment (risperidone, administered orally) plus Behavioral Intervention: "psychosocial treatment" included "psychoeducation" "social skills" "healthy life style habits" "exercise in group"
  Other Names: "Psychoeducation"; "Social Skills"; "Healthy Life style"; "Exercise in group"
  Arms: 1 Guideline treatment
Drug: Treatment as Usual (any other antipsychotic) — Participants will receive the Treatment as Usual (atypical antipsychotic) plus Behavioral Intervention: psychosocial treatment assigned by clinician.
  Other Names: Any other antipsychotic assigned by clinician
  Arms: 2 Treatment as Usual

SUMMARY:
The purpose of this study was to evaluate the applicability and usefulness of the guideline treatment for diagnosis and treatment of adolescents with schizophrenia, also to evaluate the compliance to the treatment according to the guidelines, and to compare the treatment compliance, severity of illness and social functioning of patients treated according to guideline treatment vs patients with the treatment as usual on a six month follow up.

DETAILED DESCRIPTION:
The drug treatment of patients on the Guideline Treatment group followed an algorithm, where an atypical antipsychotic must be maintained during 6 weeks before the evaluation of medication change if the PANSS score did not show a reduction of 30% and the patients did not show functional improvement. Clozapine could be administered if two trials of antipsychotics were not effective. Benzodiazepines, antidepressants, anticholinergics or anticonvulsants were allowed for the treatment of comorbid disorders or side effects.

The psychosocial treatment included psychoeducation (three 90 min sessions with the family and two 45 min sessions with the patients), followed by a seven 45 min sessions training on social skills which focused on verbal and non-verbal communication, as well as in conversation skills. Patients were also trained in healthy life style habits and were included on a 30 min of exercise in group.

TAU included an antipsychotic and the psychosocial treatment decided by the clinician

ELIGIBILITY:
Inclusion Criteria:

* Total score ≥ 70 on the Positive and Negative Syndrome Scale (PANSS) and a score of at least 4 (moderate) on 3 of the follow core items (conceptual disorganization , hallucinatory behavior, suspiciousness, and unusual thought content).
* Patients were required to have a score of ≥ 4 symptoms on the Clinical Global Impression Improvement Scale (CGI-S)
* Had not received antipsychotic in proper doses/ a regular antipsychotic treatment for at least 4 weeks previous enrollment.

Exclusion Criteria:

* Unstable medical conditions
* Their diagnosis changed during the study
* Had a history of substance dependence or substance use (except cannabis), -Females with pregnancy
* Refusal to practice contraception during the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Responder status, >30% reduction in PANSS score and improvement on CGI score. | six months
  Responder status, defined by >30% reduction in PANSS scores and significant improvement on the CGI score. CGI significant improvement defined as a score of 1 (very much improved), or 2 (much improved).

SECONDARY OUTCOMES:
Functional outcomes assessed by the Personal and Social Performance Scale. | six months
  Functional outcomes assessed by the Personal and Social Performance Scale. The lowest score represents lack of autonomy in the basic functioning and the highest score reflects excellent performance.
Cognition assessed using The MATRICS Consensus Cognitive Battery (MCCB) | six months
  Cognition assessed using "The MATRICS Consensus Cognitive Battery"; includes ten trials evaluating seven cognitive domains; processing speed, verbal learning and visual, verbal working memory and non-verbal reasoning and problem solving, sustained attention, and social cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa E. Ulloa, Md Phd, Principal Investigator — Secretaria de Salud

IPD SHARING:
Plan to Share IPD: Undecided